CLINICAL TRIAL: NCT01357226
Title: Using the Bp TRU in Clinical Settings: a Knowledge Translation Study
Brief Title: Using the Blood Pressure TRU in Clinical Settings: a Knowledge Translation Study
Status: Completed | Type: Observational
Sponsor: North Toronto Primary Care Research Network (Network)
Responsible Party: Principal Investigator, Michelle Greiver, Dr. Michelle Greiver, North Toronto Primary Care Research Network
Other Study IDs: 11-0519
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-01

CONDITIONS: Blood Pressure
Keywords: measurement in two environments

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients over the age of 18

SUMMARY:
Context: Use of automated blood pressure (BP) measurement devices in the office setting is increasingly recognized as superior to manual BP measurement. Current recommendations are to have the patient alone in a quiet room, with no interactions with health care professionals during the readings. However, this may not be practical in primary care offices where the exam rooms are constantly being used.

Objective: To compare measurements with an automated BP device in private examination rooms with measurements in non-private areas of a primary care office.

Design: Randomized controlled trial with cross-over.

Setting: Community based primary care office participating in the NorTReN Practice Based Research Network in Toronto, Ontario.

Participants: Fifty consecutive consenting patients over the age of 18 having their BP checked as part of their routine care.

Intervention: Patients will be randomly allocated to either automated BP measurement in an exam room, or in a non-private area of the clinic. After being tested in the first location they will subsequently be tested in the second location with the same device.

Main outcome measure: The primary outcome measure is a comparison between the mean systolic values of the automated BP measurements in the two office areas. The investigators will use the t-test for paired samples. The secondary outcome is a comparison of systolic values for patients with previously documented hypertension. The investigators define a clinically meaningful result as a difference of 5 mmHg or more in systolic BP.

Conclusion: New technology is more readily adopted if barriers to use are minimized. If the investigators find no differences in BP readings between office locations, physicians will then have the convenience of an additional office area to implement the automated BP measurement device.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent
* Over the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to a community-based primary care office for routine blood pressure measurement.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Automated Blood Pressure measurements in two different environments | Day of consent
  Comparison of the mean systolic values of the automated blood pressure measurement in the private exam room and the common area (laboratory area).

SECONDARY OUTCOMES:
Automated Blood Pressure values of hypertensive patients in two different environments | Day of consent
  Comparison of the mean systolic blood pressure measurements for patients with previously documented hypertension in the private exam room and the common area (laboratory area).

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Greiver, MD, Principal Investigator — North Toronto Primary Care Research Network
Locations (1):
- North York Family Health Team, North York, Ontario, Canada